CLINICAL TRIAL: NCT00726076
Title: Managing Epilepsy Well: Self-Management Intervention Research-Coordinating Center
Brief Title: Managing Epilepsy Well- WebEase Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Colleen K Diiorio, PhD, Professor Emerita, Emory University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00006628; 5 U48 DP00004304 (Other: Other)
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Epilepsy
Keywords: Epilepsy; Medication; Stress; Sleep; Lifestyle Management
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): The Treatment Group received the WebEase Intervention immediately after completing the Baseline Assessment.
  Interventions: Behavioral: WebEase
- Control (Experimental): Control Group also received the WebEase Intervention. However, Control Group participants began the Intervention 6 weeks after completing the Baseline Assessment.
  Interventions: Behavioral: WebEase

INTERVENTIONS:
Behavioral: WebEase — Computer-based epilepsy self-management program
  The Treatment Group received the WebEase Intervention immediately after completing the Baseline Assessment
  Arms: Treatment
Behavioral: WebEase — Control Group also received the WebEase Intervention. However, Control Group participants began the Intervention 6 weeks after completing the Baseline Assessment.
  Arms: Control

SUMMARY:
The purpose of this study is to test a computer program for people with epilepsy. The program was developed to help people with epilepsy improve their self-management skills for taking medications, reducing stress, and sleeping well.

DETAILED DESCRIPTION:
WebEase is an internet self-management program for people with epilepsy. Our goal is to offer a program that supports the management of epilepsy by people with epilepsy. The program is based on proven techniques of motivational interviewing and stages of change. Before offering WebEase to the general public, we tested the program among volunteers with epilepsy. We recruited individuals with epilepsy who were willing to use the program.

The program was developed by a team of researchers and physicians who treat patients with epilepsy. The program offers information on three major topics: 1) medication taking, 2) stress and 3) sleep management as it relates to epilepsy. It includes quizzes, fact sheets, and links to other authoritative websites on epilepsy.

Before beginning the study, each participant completed a brief survey about medications, stress, and sleep. Then participants worked through the WebEase program. WebEase consists of three modules: medication, stress, and sleep. Each module lasts 2 weeks, and includes an interactive session geared specifically to each person's needs. During the study, each participant kept a diary of medications, stress, sleep, and seizures, which allowed them to see changes over time. After completing the WebEase program, participants completed two more brief surveys about six weeks apart. About half of the participants were asked to complete two surveys about 6 weeks apart before beginning the WebEase program. These individuals completed one survey after the end of the program.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Understand and speak English
* Have been diagnosed with epilepsy
* Have been on an antiepileptic medication (AED) for at least 3 months
* Have access to the internet
* Be willing to participate
* Have not participated in WebEase in the past

Exclusion Criteria:

* Under age 18
* Unable to understand and speak English
* Have NOT been diagnosed with epilepsy
* Have NOT been on an AED for at least 3 months
* Not willing to participate
* Have participated in WebEase in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2008-07; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Epilepsy self-management: medication adherence, stress level, and sleep quality | Baseline- 6 weeks- 12 weeks

SECONDARY OUTCOMES:
Seizure frequency | Baseline- 6 weeks- 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Colleen DiIorio, PhD, RN, Principal Investigator — Rollins School of Public Health, Emory University
Locations (1):
- Rollins School of Public Health, Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Background] Walker ER, Bamps Y, Burdett A, Rothkopf J, Diiorio C. Social support for self-management behaviors among people with epilepsy: a content analysis of the WebEase program. Epilepsy Behav. 2012 Mar;23(3):285-90. doi: 10.1016/j.yebeh.2012.01.006. Epub 2012 Feb 23. PMID 22364762
- [Result] DiIorio C, Bamps Y, Walker ER, Escoffery C. Results of a research study evaluating WebEase, an online epilepsy self-management program. Epilepsy Behav. 2011 Nov;22(3):469-74. doi: 10.1016/j.yebeh.2011.07.030. Epub 2011 Sep 1. PMID 21889413